CLINICAL TRIAL: NCT02443012
Title: Evaluation on Efficacy of Topical Nepafenac as Supplement Therapy in the Treatment of Diabetic Macular Edema
Brief Title: Topical Nepafenac as Supplement for Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Jan Bond Chan, Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRR-13-1296-13714; 1001/PPSP/812064 (Other Grant/Funding Number: Research University Grant (USM))
Record Dates: First submitted 2015-04-25; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Nepafenac; Laser therapy; Clinically significant macular edema; Adjunct Treatment; Topical Nepafenac
MeSH Terms: interventions — nepafenac; Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nevanac (Experimental): Patients with CSME treated with argon laser photocoagulation (focal/grid laser) and Topical Gutt Nepafenac 0.1% given 8 hourly interval for 3 months
  Interventions: Drug: Topical Gutt Nepafenac 0.1%; Procedure: Laser
- Laser (Placebo Comparator): Patients with CSME treated with argon laser photocoagulation (focal/grid laser)
  Interventions: Procedure: Laser

INTERVENTIONS:
Drug: Topical Gutt Nepafenac 0.1% — Topical Nepafenac as an adjunct to focal/grid laser
  Other Names: Nevanac
  Arms: Nevanac
Procedure: Laser — Grid/Focal Laser Photocoagulation

SUMMARY:
Diabetic macular edema (DME) is a major cause of visual loss in patients with diabetes mellitus. The standard treatment is with focal/grid laser therapy. Topical nepafenac was used as an adjunct therapy for treatment of DME.

The aim of this study is to compare the difference of best corrected visual acuity (BCVA) and central macular thickness (CMT) at 3 months post treatment between combination therapy of laser and topical nepafenac and laser monotherapy in patients with DME.

DETAILED DESCRIPTION:
Diabetes mellitus with its systemic complications has been an enormous health treat to the world population today. In the US, the ophthalmic related complications has been estimated to cause up to 4.2 million (28.5%) people in 2005 till 2008 to suffer from blindness. One of the most common causes of visual acuity loss in patients with diabetes mellitus is diabetic macular edema (DME).

The gold standard of treatment for clinically significant macular edema (CSME), a form of DME, is through focal and grid laser as shown by the Early Treatment Diabetic Retinopathy Study. The development of newer drugs such as anti vascular endothelial growth factors anti (VEGFs), an alternative to laser treatment, has become a topic of interest in the recent years. Other alternative to treatment of DME is steroid such as triamcinolone injection and dexamethasone injections. However, both anti VEGFs and steroids are expensive and not readily available in all centres. Both types of medications require repeated treatment and the route of administration through intravitreal also poses risk of endophthalmitis, lens injury, retinal detachment, vitreous hemorrhage, increase in intraocular pressure and cataract.

The pathophysiology of DME is not fully understood yet. It was suggested that it is likely to be a chronic low-grade inflammation. Through this theory, topical non-steroidal anti-inflammatory drugs (NSAIDs) have been used to treat DME. The investigators postulate that the addition of topical NSAIDs in patients receiving standard treatment of laser therapy may help to improve the outcome of patients with DME. It has the advantage of no needles involved, convenient, easy to use and minimal side effects. The aim of this study is to evaluate the outcome of visual acuity and macular thickness at 3 months post treatment between laser monotherapy and combination of laser and topical nepafenac in DME.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus with CSME
* Aged 18 to 70 years old
* Clear media (Able to perform OCT)
* HbA1c less than 12% at 3 months

Exclusion Criteria:

* CSME with severe Non-Proliferative Diabetic Retinopathy (NPDR) or Proliferative Diabetic Retinopathy(PDR)
* Previous laser treatment
* Previous ocular injury or surgery
* History of taking topical or systemic anti inflammatory agents
* Allergic to NSAIDs
* Other ocular pathology (ARMD, Glaucoma, IPCV)
* High myope

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in Logarithm Best Minimal Angle of Resolution Corrected Visual Acuity (LogMAR BCVA) (Measurement of Visual Acuity) | 3 months
  Measurement of Best Corrected Visual Acuity by means of refraction using the ETDRS Chart

SECONDARY OUTCOMES:
Changes in central macular thickness (measurement of macular thickness) | 3 months
  Measurement of macular thickness using Spectralis OCT

OTHER OUTCOMES:
Safety profile of topical nepafenac as assessed by side effects (such as keratitis, eye redness and blepharitis and epithelial defect) | 3 months
  We look into side effects of topical NSAIDs such as keratitis, eye redness and blepharitis and epithelial defect.

CONTACTS AND LOCATIONS:
Overall Officials: Zunaina Embong, MS Ophthal, Study Chair — Universiti Sains Malaysia
Locations (2):
- Malaysia (2):
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Selayang, Batu Caves, Selangor

REFERENCES:
- [Background] Callanan D, Williams P. Topical nepafenac in the treatment of diabetic macular edema. Clin Ophthalmol. 2008 Dec;2(4):689-92. doi: 10.2147/opth.s3965. PMID 19668417
- [Background] Hariprasad SM, Callanan D, Gainey S, He YG, Warren K. Cystoid and diabetic macular edema treated with nepafenac 0.1%. J Ocul Pharmacol Ther. 2007 Dec;23(6):585-90. doi: 10.1089/jop.2007.0062. PMID 18001248